CLINICAL TRIAL: NCT03675906
Title: The Relationship Between Preoperative and Postoperative Hypoalbuminemia and Development of Acute Kidney Failure (AKI) According to KDIGO Criteria in Advanced Age Hip Kidney Surgery
Brief Title: The Relationship Between Hypoalbuminemia and Development of Acute Kidney Failure (AKI) According to KDIGO Criteria
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Erzincan University (Other)
Responsible Party: Principal Investigator, ILKE KUPELI, principal investigator, Erzincan University
Other Study IDs: ERZINCAN BINALI YILDIRIM
Record Dates: First submitted 2018-09-12; First posted 2018-09-18 (Actual); Last update posted 2018-09-18 (Actual); Status verified 2018-09

CONDITIONS: Hypoalbuminemia; Acute Kidney Failure
Keywords: hypoalbuminemia; Acute Kidney Failure; older age; hip fracture
MeSH Terms: conditions — Hypoalbuminemia; Acute Kidney Injury; Hip Fractures

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- preoperative albumin levels <3.8
  Interventions: Other: hypoalbuminemia
- preoperative albumin level >3.8
  Interventions: Other: hypoalbuminemia
- postoperative Day 2 albumin level <2.9
  Interventions: Other: hypoalbuminemia
- postoperative Day 2 albumin level >2.9
  Interventions: Other: hypoalbuminemia

INTERVENTIONS:
Other: hypoalbuminemia — hypoalbuminemia and acute kidney injury

SUMMARY:
This study was designed to determine the association between preoperative and postoperative hypoalbuminemia and AKI in older age hip fracture surgeons, to determine which period of hypoalbuminemia contributes more to AKI development, the incidence of AKI according to anesthesia type, the presence of other factors affecting AKI development, the duration of hospitalization and cost- to be investigated.

ELIGIBILITY:
Inclusion Criteria:

* patients with femur fracture surgery
* 65 years and over
* Patients with ASA I - IV physical condition
* patients with spinal anesthesia or peripheral nerve block

Exclusion Criteria:

* Patients undergoing emergency surgery
* patients with preoperative serum creatinine (sCr) level> 1.5 mg / dl
* patients with low serum albumin levels in both preoperative and postoperative periods
* patients receiving preoperative ventilator care
* patients with spinal anesthesia or peripheral nerve block contraindications (coagulopathies, local infection at the puncture site, spot infection) or nonsteroidal antiinflammatory drug (NSAID)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: ASA I - IV physical status and under spinal anesthesia or peripheric nerve block, 160 patients over 65 years of age undergoing femoral fracture surgery between 01.01.2018 - 01.07.2018
Sampling Method: Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2018-09-12 (Actual); Primary Completion 2018-12-15 (Estimated); Study Completion 2018-12-30 (Estimated)

PRIMARY OUTCOMES:
hypoalbuminemia and AKI - incidence of AKI | 3 months
  hypoalbuminemia and incidence of AKI according to KDIGO criterias

SECONDARY OUTCOMES:
anesthesia type - incidence of AKI | 3 months
  incidence of AKI according to anesthesia type

CONTACTS AND LOCATIONS:
Locations (1):
- Erzincan University, Erzincan, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Section 2: AKI Definition. Kidney Int Suppl (2011). 2012 Mar;2(1):19-36. doi: 10.1038/kisup.2011.32. No abstract available. PMID 25018918
- [Result] Kim HJ, Koh WU, Kim SG, Park HS, Song JG, Ro YJ, Yang HS. Early postoperative albumin level following total knee arthroplasty is associated with acute kidney injury: A retrospective analysis of 1309 consecutive patients based on kidney disease improving global outcomes criteria. Medicine (Baltimore). 2016 Aug;95(31):e4489. doi: 10.1097/MD.0000000000004489. PMID 27495094
- [Result] Kim K, Bang JY, Kim SO, Kim S, Kim JU, Song JG. Association of preoperative hypoalbuminemia with postoperative acute kidney injury in patients undergoing brain tumor surgery: a retrospective study. J Neurosurg. 2018 Apr;128(4):1115-1122. doi: 10.3171/2016.11.JNS162237. Epub 2017 May 5. PMID 28474996
- [Result] Shin KH, Han SB. Early postoperative hypoalbuminemia is a risk factor for postoperative acute kidney injury following hip fracture surgery. Injury. 2018 Aug;49(8):1572-1576. doi: 10.1016/j.injury.2018.05.001. Epub 2018 May 2. PMID 29908852